CLINICAL TRIAL: NCT04833868
Title: Efficacy of Hippotherapy Combined With Schroth Exercises on Pulmonary Function and Aerobic Capacity in Adolescents With Idiopathic Scoliosis: A Randomized Controlled Trial
Brief Title: Effect of Hippotherapy and Schroth Exercise on Pulmonary Function and Aerobic Capacity in Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Collaborators: Taif University (Other)
Responsible Party: Principal Investigator, Mohamed A. Abdel Ghafar, associate Professor, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMC
Record Dates: First submitted 2021-03-31; First posted 2021-04-06 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Scoliosis Idiopathic
Keywords: Hippotherapy; Pulmonary Function; Idiopathic Scoliosis
MeSH Terms: interventions — Equine-Assisted Therapy

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hippotherapy combined with Schroth Exercise (Experimental): received hippotherapy combined with Schroth Exercise hippotherapy session for 30 minutes of walking and sitting trot training, 15 sessions split into 2 phases over ten weeks in addition to 60-minute session Schroth's intervention, 3 times/ week for 10 weeks
  Interventions: Other: hippotherapy and schroth exercise
- Schroth Exercise (Active Comparator): received Schroth's intervention for a 60-minute session, 3 times/ week for 10 weeks
  Interventions: Other: schroth exercise

INTERVENTIONS:
Other: hippotherapy and schroth exercise — pulmonary function and aerobic capacity were measured in patients with mild idiopathic scoliosis before and after 10-week hippotherapy intervention combined with Schroth exercise
  Arms: hippotherapy combined with Schroth Exercise
Other: schroth exercise — pulmonary function and aerobic capacity were measured in patients with mild idiopathic scoliosis before and after 10-week of Schroth exercise
  Arms: Schroth Exercise

SUMMARY:
BACKGROUND: Idiopathic scoliosis has been identified as a common spinal malalignment that negatively impacts the respiratory system and physical conditioning in adolescents. Hippotherapy is an equestrian intervention that optimizes physical performance and mobility in a bunch of contexts; however, its influence on pulmonary function remains unclear.

AIM: This research aimed to analyze the impact of ten weeks of hippotherapy combined with Schroth exercises on ventilatory function and aerobic capacity in AIS.

DESIGN: Randomized Controlled Trial SETTING: Outpatients attend a single center that includes a rehabilitation room and recreational riding center.

POPULATION: Forty-five patients were arbitrarily recruited to the experimental (N= 22) and control group (N=23).

METHODS: Patients in the experimental group received 30 minutes of walking and sitting trot training, 15 sessions split into 2 phases over ten weeks. The two groups attended a 60-minute session of Schroth's intervention, 3 times/ week for 10 weeks. Two-way ANOVA for between-group comparisons and independent t-test for within-group comparisons were used in the statistical analysis.

DETAILED DESCRIPTION:
A total of 45 patients (13 males and 32 females) participated in the current study. The participants were assigned to one of two groups in a random manner: an experimental group who received hippotherapy combined with Schroth Exercise and the control group who received only schorth exercise. (FVC, FEV1, FEV1/FVC, MVV, and 6MWT) were measured before and after 10 weeks intervention

ELIGIBILITY:
Inclusion Criteria:

* all types of curves,
* curves between 10 and 20 degrees (29),
* Risser grade 0 to 5
* the availability to be engaged in once a week visit

Exclusion Criteria:

Adolescents with:

* obstructive pulmonary diseases
* associated neuromuscular diseases
* recent infectious episodes in the previous two months
* history of cardiovascular or psychological disorders
* any significant history of riding horses

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-03-07 (Actual)

PRIMARY OUTCOMES:
FVC in liters | ten weeks
  change in FVC measured Using Spiromaster PC-10 Spirometer
FEV1 in liters | ten weeks
  change in FEV1 measured Using Spiromaster PC-10 Spirometer
MVV in liters/min | ten weeks
  change in MVV measured Using Spiromaster PC-10 Spirometer
FEV1/FVC in percentage | ten weeks
  change in FEV1/FVC measured Using Spiromaster PC-10 Spirometer
aerobic capacity | ten weeks
  6MWT

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M. Abdel Ghafar, Ph.D, Principal Investigator — Batterjee Medical College
Locations (1):
- Battarjee Medical College, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No